CLINICAL TRIAL: NCT06480123
Title: Skin Drug Prepared From Stem Cell Derived Exome for Treatment of Diabetic Foot: a Phase II Clinical Trial
Brief Title: Stem Cell Derived Exome for Treatment of Diabetic Foot
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-SC-EXOME-DF 026
Record Dates: First submitted 2024-06-23; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot; Stem Cell
Keywords: Diabetic foot; Stem cell; Exome; Skin drug
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem Cell Derived Exome (Experimental)
  Interventions: Drug: Skin drug prepared with exome originated from stem cell

INTERVENTIONS:
Drug: Skin drug prepared with exome originated from stem cell — Skin drug prepared with exome originated from stem cell will be applied to patient with diabetic foot.

SUMMARY:
This trial is designed to investigate the safety and efficacy of patients with diabetic foot by using stem cell derived exome.

DETAILED DESCRIPTION:
It is estimated that about 150 million people are suffering diabetes mellitus, of whom more than 15% will develop foot ulcers or gangrene at some times, so called diabetic foot. The diabetic foot is very difficult to cure by traditional approaches.

This phase I clinical trial is designed to assess the safety and theraputical benefit of the stem cell derived exome.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of diabetic foot.
2. Signed informed consent before recruiting.
3. Age above 18 years or less than 90 years.
4. ECOG score < 4
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients have poor compliance.
5. Allergic to the skin drug;
6. Any agents which could affect the absorption or pharmacokinetics of the study drugs
7. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the treatment | Six months
  Safety will be assessed by recording all types of advise effects upon and after the treatment.
Efficacy of the treatment | Six months
  Efficacy will be defined as objective response rate + steady disease rate.

SECONDARY OUTCOMES:
Duration of remission (DOR) | 5 years
  DOR will be defined as the duration of the diabetic foot remission.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China